CLINICAL TRIAL: NCT05639972
Title: A Feasibility Study of E7 TCR-T Cell Induction Therapy for Locoregionally Advanced HPV-Associated Cancers
Brief Title: E7 T-cell Receptor (TCR) -T Cell Induction Therapy for Locoregionally Advanced HPV-associated Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Christian Hinrichs (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christian Hinrichs, Chief, Section of Cancer Immunotherapy, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192104; Pro2022000437 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: HPV-Associated Cervical Carcinoma; HPV-Related Carcinoma; HPV-Related Malignancy; HPV Positive Oropharyngeal Squamous Cell Carcinoma; HPV-Related Adenocarcinoma; HPV-Related Adenosquamous Carcinoma; HPV-Related Squamous Cell Carcinoma; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Penile Squamous Cell Carcinoma; HPV-Related Vulvar Squamous Cell Carcinoma; HPV-Related Endocervical Adenocarcinoma; Cervical Cancer; Oropharynx Cancer; Anal Cancer; Vulvar Cancer; Penile Cancer; Vaginal Cancer
Keywords: HPV; Cell therapy; Adoptive cell therapy; Immunotherapy; Radiation; Chemoradiation; CAR-T, cell therapy; Tumor infiltrating lymphocyte; TCR; T cell; Gene therapy; Cervical cancer; Oropharyngeal cancer; Anal cancer; Vulvar cancer; Vaginal cancer; Penile cancer; Induction therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Anus Neoplasms; Vulvar Neoplasms; Penile Neoplasms; Vaginal Neoplasms | interventions — Adoptive Transfer; aldesleukin

STUDY DESIGN:
Intervention Model Description: This is a single-arm feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- E7 TCR-T cells (Experimental): Subjects will receive a conditioning regimen, E7 TCR-T cells, and aldesleukin.
  Interventions: Biological: E7 TCR-T cells; Drug: Aldesleukin

INTERVENTIONS:
Biological: E7 TCR-T cells — Participants will receive a conditioning regimen consisting of cyclophosphamide and fludarabine. E7 TCR-T cells will be administered as a single intravenous infusion.
  Other Names: E7 TCR; HPV TCR; TIL; Adoptive cell transfer; CAR-T; TCR
Drug: Aldesleukin — Within 24 hours after E7 TCR-T cell infusion, aldesleukin 720,000 IU/kg IV will be administered every 8 hours as an inpatient for up to 3 doses. Aldesleukin dosing will be stopped for aldesleukin-related grade 3 or greater toxicity other than flushing, fever, chills, or hemodynamic changes (tachycardia or hypotension) that respond to crystalloid infusion. Aldesleukin may also be stopped at any time at investigator discretion.
  Other Names: Proleukin

SUMMARY:
The goal of this study is to determine the feasibility of administration of a single dose of E7 TCR-T cells as induction therapy prior to definitive treatment (chemoradiation or surgery) of locoregionally advanced HPV-associated cancers. The intent of E7 TCR-T cell treatment is to shrink or eliminate tumors and thereby facilitate definitive therapy and increase overall survival.

This study seeks to determine 1) if E7 TCR-T cells can be administered without undue delay in definitive treatment, 2) the tumor response rate to E7 TCR-T cell treatment, and 3) the disease-free survival rate at 2 and 5 years.

Participants will undergo an apheresis procedure to obtain T cells that will be genetically engineered to generate E7 TCR-T cells. They will receive a conditioning regimen, a single infusion of their own E7 TCR-T cells, and adjuvant aldesleukin. Participants will follow up to assess safety and determine tumor response and will return to their primary oncology team for definitive therapy.

DETAILED DESCRIPTION:
This is a single-arm, single-cohort, single-center, feasibility study to determine the feasibility of E7 TCR-T cell induction therapy for locoregionally advanced human papillomavirus (HPV)-associated cancers (LAHPVC). Participants must have LAHPVC with HPV-16-positive cancer (tumor test) and the human leukocyte antigens (HLA)-A*02:01 allele (blood test). Participants will undergo apheresis for generation of autologous, gene-engineered, E7 TCR-T cells. One week after apheresis, they will receive a non-myeloablative lymphocyte-depleting preparative regimen of cyclophosphamide and fludarabine. Conditioning will be followed by a single infusion of E7 TCR T cells and adjuvant high-dose aldesleukin. Participants will follow up 3 weeks and 6 weeks after treatment. Tumor response will be assessed by imaging studies at the 6-week time point. Participants will be referred back to their primary oncology team for definitive therapy after the 6-week assessment (or earlier if tumors do not appear to be responding). Participants will be followed to determine 2- and 5-year disease free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed carcinoma of a primary tumor site and stage indicated in Table 3 of the protocol.
2. Tumor with HPV16 genotype as determined by testing performed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory.
3. HLA-A*02:01 allele determined by testing performed in a CLIA certified laboratory. Participants may be enrolled based on low resolution typing (i.e., HLA-A*02) but the HLA-A*02:01 allele type must be confirmed prior to apheresis.
4. Measurable disease per RECIST Criteria Version 1.1 or PERCIST.
5. Age > 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
7. Negative pregnancy test for women under 55 and all women who have had a menstrual period in the last 12 months. A pregnancy tests is not required for women who have had a bilateral oophorectomy or hysterectomy.
8. Men and women of child-bearing potential must agree to use adequate contraception (i.e., intrauterine device, hormonal barrier method of birth control; abstinence; tubal ligation or vasectomy) prior to study entry and for four months after treatment. Should a women become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
9. Seronegative for HIV antibody, hepatitis B surface antigen (sAg), and hepatitis C antibody. If a hepatitis C antibody test is positive, then testing for antigen by reverse transcription polymerase chain reaction (RT-PCR) must be negative.
10. Participants must have organ and marrow function as defined below:

    1. Leukocytes > 3,000/Mantle cell lymphoma (mcL)
    2. Absolute neutrophil count > 1,500/mcL
    3. Platelets > 100,000/mcL
    4. Hemoglobin > 9.0 g/dL
    5. Total bilirubin within normal institutional limits except in participants with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL.
    6. Serum aspartate aminotransferase (AST) (SGOT)/ alanine transaminase (ALT)(SGPT) < 2.5 x upper limit of normal (ULN)
    7. Calculated creatinine clearance (CrCl) >50 mL/min/1.73 m2for participants with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation).
    8. international normalized ratio (INR) or activated partial thromboplastin time ( aPTT) ≤1.5 X ULN unless the subject is receiving anticoagulant therapy. Subjects on anticoagulant therapy must have a PT or aPTT within therapeutic range and no history of severe hemorrhage.
11. Participants must be able to understand and be willing to sign the written informed consent document.
12. Participants must agree to participate in protocol CINJ 192103 (Pro2021002307) for gene therapy long term follow up and in protocol Cancer Institute of New Jersey (CINJ) 192002 (Pro2021000281) for biospecimen collection study.

Note: Patients may have undergone minor surgical procedures with the past three weeks, as long as all toxicities have recovered to Grade 1 or less.

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participation in this study:

1. Prior systemic therapy or definitive chemoradiation for the cancer that is being treated on this protocol.
2. Current treatment with another investigational agent.
3. History of severe allergic reactions to compounds of similar chemical or biological composition to agents used in this study.
4. Uncontrolled intercurrent illness such as active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
5. Subjects with HLA-A*02:01 damaging mutation or allele loss or other molecular resistance detected by research or clinical sequencing will not be eligible.
6. Documented LVEF of less than or equal to 45% tested. The following participants will undergo cardiac evaluations:

   1. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or
   2. Age > 50 years old
7. Participants with baseline screening pulse oxygen level of <92% on room air will not be eligible. If the underlying cause of hypoxia improves, they may be reevaluated.
8. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T cells, breastfeeding should be discontinued if the mother is treated with E7 TCR T cells. These potential risks may also apply to other agents used in this study.
9. Participants with a systemic immunodeficiency including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Participants who have decreased immune competence may be less responsive to the treatment.
10. Participants on immunosuppressive drugs including corticosteroids unless meeting criteria outlined in Section 6.1 (Prohibited Medications).
11. Participants with potentially severe autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis, autoimmune pancreatitis, or systemic lupus erythematosus are not eligible. Patients with less severe autoimmune diseases such as hypothyroidism, vitiligo, and other minor autoimmune disorders are eligible.
12. Participants with prior or concurrent malignancy whose natural history or treatment is unlikely to interfere with the safety or efficacy assessments of the investigational regimen are eligible for this trial. Examples include, but are not limited to:

    1. Carcinoma in situ
    2. Cutaneous skin cancers requiring only local excision
    3. Low grade non-muscle invasive bladder cancer
    4. Low grade prostate cancer
13. Subjects who received a live vaccine within 30 days prior to enrollment are not eligible.
14. Determination by the Principal Investigator that participation is not in the best interest of the research subject or may jeopardize the safety of the subject or integrity of the clinical trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of administering E7 TCR-T cell therapy as induction treatment for LAHPVC | 6 weeks
  Proportion of subjects who complete treatment without an event that meets criteria for feasibility failure

SECONDARY OUTCOMES:
Objective tumor response rate at 6-weeks after treatment | 6 weeks
  Tumor response as assessed by imaging using Response Evaluation Criteria in Solid Tumors (RECIST) criteria Version 1.1 or PERCIST
2-year and 5-year disease free survival (DFS) | 5 years
  DFS will be determined using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Data will be made available through the publisher at the time of publication.
Access Criteria: Data will be accessible through the publisher.

REFERENCES:
- [Background] Nagarsheth NB, Norberg SM, Sinkoe AL, Adhikary S, Meyer TJ, Lack JB, Warner AC, Schweitzer C, Doran SL, Korrapati S, Stevanovic S, Trimble CL, Kanakry JA, Bagheri MH, Ferraro E, Astrow SH, Bot A, Faquin WC, Stroncek D, Gkitsas N, Highfill S, Hinrichs CS. TCR-engineered T cells targeting E7 for patients with metastatic HPV-associated epithelial cancers. Nat Med. 2021 Mar;27(3):419-425. doi: 10.1038/s41591-020-01225-1. Epub 2021 Feb 8. PMID 33558725